CLINICAL TRIAL: NCT05782166
Title: Cross-Cultural Adaptation of a Betel Quid Cessation Program and Evaluation of Its Effectiveness in a Malaysian High-Risk Community
Brief Title: Adapting a Betel Quid Cessation Program for a High-risk Community in Malaysia and Evaluating Its Effectiveness
Acronym: M-BENIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Collaborators: University of Hawaii Cancer Research Center (Other); University of Guam (Other)
Responsible Party: Principal Investigator, Mary Melissa A/P Sarimuthu, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSCH ID-23-00412-TVU
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Betel Nut Chewer; Tobacco Cessation
Keywords: Betel Quid; Cessation Program; Effectiveness
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Betel Quid Cessation via Educational Booklet (Placebo Comparator): Participants will be given only an educational booklet on screening day (Day-1) and will be followed up on Day-22 and Month-3 to assess their current chewing status and other related parameters.
  Interventions: Behavioral: Betel Quid Educational Booklet
- Betel Quid Cessation via Educational Booklet & Intervention Module (Experimental): Participants will undergo a 5-intervention sessions which will enhance their self-efficacy o quit their chewing behaviour. During the intervention sessions, they will be guided on how to monitor their chewing triggers, the lifestyle changes that they can potentially make, how to tap on their social support system to aid in their cessation efforts and others. The intervention will last for 22 days and a follow-up session will be made on Month-3.
  Interventions: Behavioral: Betel Quid Educational Booklet; Behavioral: Betel Quid Cessation Intervention Module

INTERVENTIONS:
Behavioral: Betel Quid Educational Booklet — Eligible and consented participants will be interviewed for baseline questionnaire completion. Details regarding participants' demographics, betel quid chewing behaviours, betel quid composition, betel quid dependency levels, reasons for chewing, readiness and self-perceived barriers to quit will be obtained. Saliva samples will be obtained.
  Participants will be given an educational booklet containing general information regarding betel quid and areca nut, risk associated with betel quid chewing behaviour, cessation strategies that are modeled after tobacco cessation and some relevant researcher's contact details.
  Participants will be followed up at Day-22 and Month-3 for information regarding compliance, current chewing status, number of habit cut-down (quid/day), total number of sessions attended and current betel quid composition. Saliva samples will be taken during follow-ups for the cessation verification of participant's chewing behaviour.
Behavioral: Betel Quid Cessation Intervention Module — All eligible and consented participants will be interviewed for baseline questionnaire completion. Details regarding participants' demographics, betel quid chewing behaviours, betel quid composition, betel quid dependency levels, reasons for chewing, readiness and self-perceived barriers to quit will be obtained. Saliva samples will be obtained.
  An interactive, educational talk will be given regarding the content of the educational booklet.
  Participants will undergo a 5-intervention sessions cessation program (M-BENIT) and will be given topical worksheets on every session to monitor their triggers, lifestyle changes, social support system and others.
  Participants will be followed up at Day-22 and Month-3 for information regarding compliance, current chewing status, number of habit cut-down (quid/day), total number of sessions attended and current betel quid composition. Saliva samples will be taken during follow-ups for the cessation verification of participant's chewing behaviour.
  Arms: Betel Quid Cessation via Educational Booklet & Intervention Module

SUMMARY:
The practice of betel quid chewing is known as the top 3 causes of oral cancers in Malaysia. The devastating part among Malaysians are that more than 50% of these cancer patients present at a later stage of this disease necessitating a massive surgical procedure and a costly oncological treatment to remove the tumour and restore the vital structures in the head and neck regions of the patients. In 2010, World Health Organisation recognised that the users of betel quid are having a 'Dependency Syndrome' similar to that of a cigarette smoking. Since then, much research has been focussed upon the 'addictive nature' and the cessation of this ill-health behaviour.

Malaysia's current plight is its strikingly high prevalence of betel quid users within its high-risk communities. The other challenge is the widely scattered high-risk communities across the diverse geography, locality, ethnicity, culture and native languages across the country that make cessation not an easy task but an uphill battle.

The latest available report in 2011 showed that the females in Sabah and Sarawak's indigenous communities presented with a prevalence of 28.4% being current chewers. This prevalence was way greater than the global prevalence of 10-20% of betel quid chewers reported worldwide. The female predominance among the betel quid users in Malaysia is another matter of concern as studies had claimed that females are less likely to cease chewing habit compared to their male counterparts.

Fortunately, in 2015, a feasibility study was conducted to adapt an intensive smoking cessation intervention to cater for betel quid chewers which received a high cessation rate of 65%. Later in 2018, researchers incorporated a saliva test to assess the effectiveness of a group-based intensive betel quid cessation program which also yielded a high cessation rate of 38% among the participants.

Since there is no existing betel quid cessation intervention in Malaysia, this study aims to adapt a betel quid cessation program for a high-risk community in Malaysia.

This study hypothesised that the intervention group will produce a significantly greater cessation rate compared to the control group at the 3-months follow-up assessment.

DETAILED DESCRIPTION:
1. Framework of the Intervention:

   This study will utilise a Cognitive Behavioural Therapy (CBT) framework as study showed that CBT framework yielded better success rates in betel quid cessation compared to a Basic Health Education talk or module alone. CBT provided education, encouragement, support and equipped participants with coping skills which was repeated and emphasized at every follow-up.

   The cognitive component tackles the chewer's attitude and health beliefs by educating the participants on the carcinogenicity of betel quid. Study revealed that betel quid chewers underestimated the deleterious health effects contributed by their chewing behaviour.

   The behaviour component targets to enhance participant's self-efficacy by substituting their chewing-promoting behaviours to behaviours which are more conducive to quitting. This involves identifying and managing chewing triggers, making supportive lifestyle changes and preparing social situation responses in advance to manage peer or social event pressures.

   BENIT intervention was selected as the intervention-of-choice to be cross-culturally adapted in Malaysia due to few reasons. Firstly, it was the first intervention that targets primarily the users of areca nut in an indigenous population which was similar to the study population of the high-risk groups in Malaysia. Most chewers in Malaysia chew areca nut singly and does not incorporate smokeless tobacco into their quid preparation. Secondly, the tropical marine climate of Guam Island was similar to the study site in Malaysia (Kota Belud, Sabah). Thirdly, the age of the chewers in Malaysia were mostly 40 years of age and above, thus BENIT was more appropriate to be adapted in Malaysia. Even though there was peer-led betel quid cessation intervention in Pakistan, it was not chosen as it targeted adolescent population in the school setting.
2. Research Design:

   This is a comparative prospective community trial which utilises a cluster-randomised controlled trial design involving a Bajau indigenous community in Sabah, Malaysia with a 1:1 allocation ratio. The clusters are Bajau villages that practises betel quid chewing habits in Kota Belud district in Sabah. The Bajau villages are the unit of randomisation. There are 39 Bajau villages in Kota Belud, Sabah. The eligible villages will be randomised into intervention and control groups based on the required sample size (46 participants in each arm). The intervention group will receive an educational booklet and a structured betel quid intervention program. The control group will only receive an educational booklet.
3. Research Methodology

There will be 3 phases involved in the conduct of this study.

3.1 Phase 1 : Adaptation, Validation and Translation of the Questionnaire, Educational Booklet and Intervention Module

Three components from the BENIT intervention will undergo the cross-cultural adaptation process; namely the baseline and follow-up questionnaire, educational booklet and intervention module. The adapted material will be face validated by study investigators and content validated by smoking cessation experts from Department of Social and Preventive Medicine and Centre of Addiction Science, Universiti Malaya. The validated materials will undergo forward and backward translation to the target language 'Bahasa Melayu' by bilingual linguistic experts.

3.2 Phase 2 : Pretest and Pilot test of the study

The forward translated materials will then be pretested among 8-10 participants from a Bajau community in Kota Belud, Sabah, which will not be selected as the sample of the field study to ensure the clarity and non-ambiguity of the translated material to both the interviewer and subject in terms of conceptual and operational equivalence. A subsequent pilot test will be done on the pretested material to assess its feasibility and its psychometric properties.

3.3 Phase 3 : Implementation of the study (Field Work)

A two-days training will be conducted by the principal investigator for the study facilitators who will be involved as questionnaire and worksheet interviewers and verbal translators for this study. A simulation session will be planned to practically expose the facilitators to the order and details of the intervention and study.

Prior to the start of the intervention, a promotional initiative will be conducted with the village heads 3 weeks before the implementation of the study to provide knowledge and to convince the village heads regarding the ill effects of the chewing habit to encourage his villagers to participate in the cessation program.

3.3.3 Implementation of the Study

Control group A community screening program will be organised to recruit the eligible participants. Participants will be required to provide consent, complete a baseline questionnaire through a face-to-face interview and to provide saliva sample on Day-1. An educational booklet will be provided to participants on the same day. On Day-22 and Month-3, participants are required to return to complete a follow-up questionnaire and provide saliva sample for assessment.

Intervention Group A community screening program will be organised to recruit the eligible participants. Participants will be required to provide consent, complete a baseline questionnaire through a face-to-face interview and to provide saliva sample on Day-0. An educational booklet will be provided to participants on the same day.

On Day-1 (Session 1), a brief talk will be given regarding the nature of intervention in which participants will undergo 5 sessions of support group designed to assist them to quit betel quid chewing habit over the next 22 days. Each session will take approximately 1-2 hours. An educational talk will be delivered focussing in a more detailed manner on the topics covered in the educational booklets. Participants will later be introduced to three topical worksheets; Trigger Monitoring Logs, Trigger Management Logs and Arecoline Fading Worksheet.

On Day-8 (Session 2), a summary of the triggers experienced by the participants within that community (village) will be gathered and potential strategies to manage those triggers will be discussed with the participants. Participants will be briefed that quitting chewing behaviour is more than cutting down the betel quid numbers per day or antagonising the chewing triggers. A lifestyle change is very pertinent in making an ex-chewer remain abstinent. Strategies such as lifestyle changes, excuses to reject chew invites and usage of fake chew objects will be taught to participants to empower them to manage their triggers. Two worksheets will be introduced to the participants; Non-chewing Game Plan Worksheet and Coping with High Risk Situation Worksheet. At the end of Session 2, participants will be reminded of the quit day that will be on morning of Day 15 (Session 3).

On Day-15 (Session 3), it will be the quit date for the participants. Discussion regarding potential withdrawal symptoms post-quitting and withdrawal coping strategies will be held. A Social Support for No Betel Quid Chewing Worksheet will be introduced. This worksheet is a tool to maximise the social support of the participant to quit the behaviour. Social support can be a good source of motivation and may also act as a buffer in stressful situations. Thus, they play a positive role in the success of participants in remaining abstinent of their chewing behaviour.

On Day-18 (Session 4), discussion on the overall quitting experience of the participants will be held and the negative health effects of betel quid chewing will be emphasized. Additional coping strategies will be discussed to address newer urges to chew. Reinforcement will be given for both quitters and current chewers through a talk by the principal investigator.

On Day-22 (Session 5), a follow-up questionnaire will be completed. A discussion on the overall quitting experience will be held. Strategies for Managing Thoughts worksheet will be introduced. This is a strategy to manage the thoughts that participants might have throughout their quitting journey. This method is based on the notion that mood is related to the balance of the positive and negative thoughts. When negative thoughts outweighed the positive thoughts, the result is a depressive, anxious, angry or other symptoms that may precipitate the behaviour of a risk habit such as chewing to come through. At the end of session 5, participant's saliva samples will be collected for assessment.

On Follow up Month-3, participants will return for another follow-up questionnaire completion and for the final saliva sample collection.

Saliva Sample Collection :

An amount of 1 - 2 mL saliva sample will be collected during assessment by the principal investigator via 'passive drool' method with a 20 mL length, conical shaped polypropylene tubes and initially stored at -20◦C after collection in an insulated cooler box with reusable ice packs. The principal investigator will transport the biospecimen to the Biotechnology Research Institute (BRI), Universiti Malaysia Sabah (UMS), Sabah, Malaysia. Upon arrival to the lab, it should be stored at -80 ◦C until analysis is done.

Saliva Sample Analysis :

The Liquid Chromatography-Mass Spectrometry (LCMS) analysis will be run by staff at the Biotechnology Research Institute (BRI), Universiti Malaysia Sabah (UMS). The BRI lab is located at Kota Kinabalu, Sabah which is about 1 to 1.5 hours from the study site and precaution will be taken to deliver samples within 8 hours after collection due to the quick disappearance property of areca nut biomarkers after 8 hours of collection.

ELIGIBILITY:
Inclusion Criteria:

1. A self-reported betel quid chewer who has been practising chewing habit for the past 6 months with atleast 2-3 chewing episodes per week. The ingredient of betel quid must include areca nut without or without smokeless tobacco.
2. Other optional ingredients such as inclusion of slaked lime and betel leaf in the betel quid are allowed.
3. Age of participant must be 18 years old and above
4. Participants must be residing in study location (Kota Belud, Sabah)
5. Ability to comprehend, converse and read in Bahasa Melayu and their local language (Bajau)
6. Participants who are able to provide written consent and agree to comply with all protocol-specified procedures such as providing saliva samples, participating in five 1-2 hours sessions of intervention over 22 days and agree to attend follow-up session on the third month

Exclusion Criteria:

1. Non-Malaysian citizen
2. Participants who are not willing to quit the betel quid chewing habit at the time of the study
3. Women chewers who are pregnant or nursing at the time of study
4. Individuals with psychiatric illness or special social situations that would limit their compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of participants who self-reported that they had quitted betel quid chewing behaviour from baseline at Day-22 | Day-22
  A follow-up questionnaire will be used to assess the self-reported cessation rate. This rate will represent the immediate cessation prevalence after the program
Change in the number of participants who self-reported that they had quitted betel quid chewing behaviour from baseline at Month-3 | Month-3
  A follow-up questionnaire will be used to assess the self-reported cessation rate. This rate will represent the intermediate-term cessation prevalence of the program

SECONDARY OUTCOMES:
Change in the levels of areca nut biomarkers in the saliva sample from baseline at Day-22 | Day-22
  Liquid chromatography mass spectrometry analysis will be done to the saliva samples to assess the level of arena nut biomarkers.
  Participant's areca nut biomarker levels will be compared to a standard cut-off levels; arecoline (60 ng/mL), arecaidine (10 ng/mL), guvacoline (20 ng/mL), and guvacine (6 ng/mL).
  Biomarkers level below this cut-off points represent that participants had ceased the chewing habit.
Change in the levels of areca nut biomarkers in the saliva sample from baseline at Month-3 | Month-3
  Liquid chromatography mass spectrometry analysis will be done to the saliva samples to assess the level of arena nut biomarkers.
  Participant's areca nut biomarker levels will be compared to a standard cut-off levels; arecoline (60 ng/mL), arecaidine (10 ng/mL), guvacoline (20 ng/mL), and guvacine (6 ng/mL).
  Biomarkers level below this cut-off points represent that participants had ceased the chewing habit.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Geraldine Doss, PhD, Study Chair — Universiti Malaya; Amer Siddiq Amer Nordin, PhD, Study Director — Universiti Malaya; Mary Melissa Sarimuthu, MCOH, Principal Investigator — Universiti Malaya
Locations (1):
- State Dental Health Department, Kota Kinabalu, Sabah, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Rmalli SW, Jenkins RO, Haris PI. Betel quid chewing elevates human exposure to arsenic, cadmium and lead. J Hazard Mater. 2011 Jun 15;190(1-3):69-74. doi: 10.1016/j.jhazmat.2011.02.068. Epub 2011 Feb 26. PMID 21440366
- [Background] Asthana S, Greig NH, Holloway HW, Raffaele KC, Berardi A, Schapiro MB, Rapoport SI, Soncrant TT. Clinical pharmacokinetics of arecoline in subjects with Alzheimer's disease. Clin Pharmacol Ther. 1996 Sep;60(3):276-82. doi: 10.1016/S0009-9236(96)90054-5. PMID 8841150
- [Background] Barker DJ. Fetal origins of coronary heart disease. BMJ. 1995 Jul 15;311(6998):171-4. doi: 10.1136/bmj.311.6998.171. PMID 7613432
- [Background] Chatterjee A, Deb S. Genotoxic effect of arecoline given either by the peritoneal or oral route in murine bone marrow cells and the influence of N-acetylcysteine. Cancer Lett. 1999 May 3;139(1):23-31. doi: 10.1016/s0304-3835(98)00364-4. PMID 10408905
- [Background] Bhat SJ, Blank MD, Balster RL, Nichter M, Nichter M. Areca nut dependence among chewers in a South Indian community who do not also use tobacco. Addiction. 2010 Jul;105(7):1303-10. doi: 10.1111/j.1360-0443.2010.02952.x. PMID 20642513
- [Background] Boucher BJ, Ewen SW, Stowers JM. Betel nut (Areca catechu) consumption and the induction of glucose intolerance in adult CD1 mice and in their F1 and F2 offspring. Diabetologia. 1994 Jan;37(1):49-55. doi: 10.1007/BF00428777. PMID 8150230
- [Background] Brown, R. A. (2003). Intensive behavioral treatment. The tobacco dependence treatment handbook: A guide to best practices, 118-177.
- [Background] Das A, Orlan E, Duncan K, Thomas H, Ndumele A, Ilbawi A, Parascandola M. Areca Nut and Betel Quid Control Interventions: Halting the Epidemic. Subst Use Misuse. 2020;55(9):1552-1559. doi: 10.1080/10826084.2019.1686022. PMID 32569544
- [Background] Deng JF, Ger J, Tsai WJ, Kao WF, Yang CC. Acute toxicities of betel nut: rare but probably overlooked events. J Toxicol Clin Toxicol. 2001;39(4):355-60. doi: 10.1081/clt-100105155. PMID 11527229
- [Background] Franke AA, Mendez AJ, Lai JF, Arat-Cabading C, Li X, Custer LJ. Composition of betel specific chemicals in saliva during betel chewing for the identification of biomarkers. Food Chem Toxicol. 2015 Jun;80:241-246. doi: 10.1016/j.fct.2015.03.012. Epub 2015 Mar 19. PMID 25797484
- [Background] Franke AA, Li X, Lai JF. Pilot study of the pharmacokinetics of betel nut and betel quid biomarkers in saliva, urine, and hair of betel consumers. Drug Test Anal. 2016 Oct;8(10):1095-1099. doi: 10.1002/dta.1912. Epub 2015 Dec 1. PMID 26619803
- [Background] Franke AA, Li X, Herzog TA, Paulino YC, Badowski G, Wilkens LR, Lai JF. Salivary Areca and tobacco alkaloids for bioverification in the Betel Nut Intervention Trial. Drug Test Anal. 2023 Jan;15(1):58-65. doi: 10.1002/dta.3364. Epub 2022 Oct 2. PMID 36057968
- [Background] Ghani WM, Razak IA, Yang YH, Talib NA, Ikeda N, Axell T, Gupta PC, Handa Y, Abdullah N, Zain RB. Factors affecting commencement and cessation of betel quid chewing behaviour in Malaysian adults. BMC Public Health. 2011 Feb 7;11:82. doi: 10.1186/1471-2458-11-82. PMID 21294919
- [Background] Giri S, Idle JR, Chen C, Zabriskie TM, Krausz KW, Gonzalez FJ. A metabolomic approach to the metabolism of the areca nut alkaloids arecoline and arecaidine in the mouse. Chem Res Toxicol. 2006 Jun;19(6):818-27. doi: 10.1021/tx0600402. PMID 16780361
- [Background] Guidelines Primary Prevention and Early Detection of Oral Potentially Malignant Disorders and Oral Cancers. (2018). Oral Health Program Ministry of Health Malaysia.
- [Background] Gupta PC, Warnakulasuriya S. Global epidemiology of areca nut usage. Addict Biol. 2002 Jan;7(1):77-83. doi: 10.1080/13556210020091437. PMID 11900626
- [Background] Hahn S, Puffer S, Torgerson DJ, Watson J. Methodological bias in cluster randomised trials. BMC Med Res Methodol. 2005 Mar 2;5:10. doi: 10.1186/1471-2288-5-10. PMID 15743523
- [Background] Herzog TA, Murphy KL, Little MA, Suguitan GS, Pokhrel P, Kawamoto CT. The Betel Quid Dependence Scale: replication and extension in a Guamanian sample. Drug Alcohol Depend. 2014 May 1;138:154-60. doi: 10.1016/j.drugalcdep.2014.02.022. Epub 2014 Feb 26. PMID 24629627
- [Background] Herzog, T. A, Zain, R. B, Ghani WN et al. (2014). Betel quid chewing (BQC) cessation multi-country study: Malaysia. [Unpublished manuscript].
- [Background] Herzog, T. A. (2022). Betel Nut Research in the Pacific [PowerPoint slides]. University of Hawai'i Cancer Center Honolulu, Hawai'i, USA.
- [Background] Huang, J. L., & McLeish, M. J. (1989). High-performance liquid chromatographic determination of the alkaloids in betel nut. Journal of Chromatography A, 475(2), 447-450.
- [Background] Hung DZ, Deng JF. Acute myocardial infarction temporally related to betel nut chewing. Vet Hum Toxicol. 1998 Feb;40(1):25-8. PMID 9467205
- [Background] Hung CR. Effect of lysozyme chloride on betel quid chewing aggravated gastric oxidative stress and hemorrhagic ulcer in diabetic rats. World J Gastroenterol. 2005 Oct 7;11(37):5853-8. doi: 10.3748/wjg.v11.i37.5853. PMID 16270397
- [Background] Jeng JH, Kuo ML, Hahn LJ, Kuo MY. Genotoxic and non-genotoxic effects of betel quid ingredients on oral mucosal fibroblasts in vitro. J Dent Res. 1994 May;73(5):1043-9. doi: 10.1177/00220345940730050501. PMID 8006230
- [Background] Javed F, Chotai M, Mehmood A, Almas K. Oral mucosal disorders associated with habitual gutka usage: a review. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Jun;109(6):857-64. doi: 10.1016/j.tripleo.2009.12.038. Epub 2010 Apr 9. PMID 20382045
- [Background] Kuo MY, Jeng JH, Chiang CP, Hahn LJ. Mutations of Ki-ras oncogene codon 12 in betel quid chewing-related human oral squamous cell carcinoma in Taiwan. J Oral Pathol Med. 1994 Feb;23(2):70-4. doi: 10.1111/j.1600-0714.1994.tb00259.x. PMID 8164156
- [Background] Lee CH, Lee JM, Wu DC, Hsu HK, Kao EL, Huang HL, Wang TN, Huang MC, Wu MT. Independent and combined effects of alcohol intake, tobacco smoking and betel quid chewing on the risk of esophageal cancer in Taiwan. Int J Cancer. 2005 Jan 20;113(3):475-82. doi: 10.1002/ijc.20619. PMID 15455377
- [Background] Lee CH, Ko AM, Yen CF, Chu KS, Gao YJ, Warnakulasuriya S, Sunarjo, Ibrahim SO, Zain RB, Patrick WK, Ko YC. Betel-quid dependence and oral potentially malignant disorders in six Asian countries. Br J Psychiatry. 2012 Nov;201(5):383-91. doi: 10.1192/bjp.bp.111.107961. Epub 2012 Sep 20. PMID 22995631
- [Background] Lee CY, Chang CS, Shieh TY, Chang YY. Development and validation of a self-rating scale for betel quid chewers based on a male-prisoner population in Taiwan: the Betel Quid Dependence Scale. Drug Alcohol Depend. 2012 Feb 1;121(1-2):18-22. doi: 10.1016/j.drugalcdep.2011.07.027. Epub 2011 Sep 28. PMID 21955360
- [Background] Lin SK, Chang YJ, Ryu SJ, Chu NS. Cerebral hemodynamic responses to betel chewing: a Doppler study. Clin Neuropharmacol. 2002 Sep-Oct;25(5):244-50. doi: 10.1097/00002826-200209000-00003. PMID 12410054
- [Background] Little, M. A., & Papke, R. L. (2015). Betel, the orphan addiction. J Addict Res Ther, 6(3), 130-132.
- [Background] Lopez-Vilchez MA, Seidel V, Farre M, Garcia-Algar O, Pichini S, Mur A. Areca-nut abuse and neonatal withdrawal syndrome. Pediatrics. 2006 Jan;117(1):e129-31. doi: 10.1542/peds.2005-0281. Epub 2005 Dec 15. PMID 16361222
- [Background] Lu CT, Yen YY, Ho CS, Ko YC, Tsai CC, Hsieh CC, Lan SJ. A case-control study of oral cancer in Changhua County, Taiwan. J Oral Pathol Med. 1996 May;25(5):245-8. doi: 10.1111/j.1600-0714.1996.tb01379.x. PMID 8835822
- [Background] Maling TH & Doss JG. (2016). The impact of an intervention programme on oral cancer awareness, health beliefs and practice of preventive behaviour in high-risk Sarawakian indigenous communities. [Doctoral dissertation, Universiti Malaya]
- [Background] Mall ASK, Bhagyalaxmi A. An Informal School-based, Peer-led Intervention for Prevention of Tobacco Consumption in Adolescence: A Cluster Randomized Trial in Rural Gandhinagar. Indian J Community Med. 2017 Jul-Sep;42(3):143-146. doi: 10.4103/ijcm.IJCM_25_16. PMID 28852276
- [Background] Marewski JN, Gigerenzer G. Heuristic decision making in medicine. Dialogues Clin Neurosci. 2012 Mar;14(1):77-89. doi: 10.31887/DCNS.2012.14.1/jmarewski. PMID 22577307
- [Background] Miles, D. (2019). ARTICLE:
- [Background] Lee CH, Ko AM, Warnakulasuriya S, Yin BL, Sunarjo, Zain RB, Ibrahim SO, Liu ZW, Li WH, Zhang SS, Kuntoro, Utomo B, Rajapakse PS, Warusavithana SA, Razak IA, Abdullah N, Shrestha P, Kwan AL, Shieh TY, Chen MK, Ko YC. Intercountry prevalences and practices of betel-quid use in south, southeast and eastern Asia regions and associated oral preneoplastic disorders: an international collaborative study by Asian betel-quid consortium of south and east Asia. Int J Cancer. 2011 Oct 1;129(7):1741-51. doi: 10.1002/ijc.25809. Epub 2011 Mar 8. PMID 21128235
- [Background] Moore G, Campbell M, Copeland L, Craig P, Movsisyan A, Hoddinott P, Littlecott H, O'Cathain A, Pfadenhauer L, Rehfuess E, Segrott J, Hawe P, Kee F, Couturiaux D, Hallingberg B, Evans R. Adapting interventions to new contexts-the ADAPT guidance. BMJ. 2021 Aug 3;374:n1679. doi: 10.1136/bmj.n1679. PMID 34344699
- [Background] Moss J, Kawamoto C, Pokhrel P, Paulino Y, Herzog T. Developing a Betel Quid Cessation Program on the Island of Guam. Pac Asia Inq. 2015 Fall;6(1):144-150. PMID 27057560
- [Background] Murphy KL, Liu M, Herzog TA. The Reasons for Betel Quid Chewing Scale (RBCS) for Ex-Chewers: Assessment of Factor Structure, Reliability, Validity and Measurement Invariance across Gender in a Guamanian Sample. Subst Use Misuse. 2022;57(4):522-530. doi: 10.1080/10826084.2021.2019781. Epub 2022 Jan 22. PMID 35067173
- [Background] Nair J, Ohshima H, Friesen M, Croisy A, Bhide SV, Bartsch H. Tobacco-specific and betel nut-specific N-nitroso compounds: occurrence in saliva and urine of betel quid chewers and formation in vitro by nitrosation of betel quid. Carcinogenesis. 1985 Feb;6(2):295-303. doi: 10.1093/carcin/6.2.295. PMID 3971493
- [Background] National Institutes of Health (NIH), United States Department of Health and Human Services (2022, July 14). Research Methods Resources. Parallel Group- or Cluster-Randomized Trials (GRTs). https://researchmethodsresources.nih.gov/methods/grt
- [Background] Ogunkolade WB, Boucher BJ, Bustin SA, Burrin JM, Noonan K, Mannan N, Hitman GA. Vitamin D metabolism in peripheral blood mononuclear cells is influenced by chewing "betel nut" (Areca catechu) and vitamin D status. J Clin Endocrinol Metab. 2006 Jul;91(7):2612-7. doi: 10.1210/jc.2005-2750. Epub 2006 May 2. PMID 16670168
- [Background] Pankaj, C. (2010). Areca nut or betel nut control is mandatory if India wants to reduce the burden of cancer especially cancer of the oral cavity. Int J Head Neck Surg, 1(1), 17-20.
- [Background] Papke RL, Hatsukami DK, Herzog TA. Betel Quid, Health, and Addiction. Subst Use Misuse. 2020;55(9):1528-1532. doi: 10.1080/10826084.2019.1666147. No abstract available. PMID 32569542
- [Background] Park YB, Jeon SM, Byun SJ, Kim HS, Choi MS. Absorption of intestinal free cholesterol is lowered by supplementation of Areca catechu L. extract in rats. Life Sci. 2002 Mar 8;70(16):1849-59. doi: 10.1016/s0024-3205(02)01485-6. PMID 12005171
- [Background] Paulino YC, Wilkens LR, Sotto PP, Franke AA, Kawamoto CT, Chennaux JSN, Mendez AJ, Tenorio LF, Badowski G, Pokhrel P, Herzog TA. Rationale and design of a randomized, controlled, superiority trial on areca nut/betel quid cessation: The Betel Nut Intervention Trial (BENIT). Contemp Clin Trials Commun. 2020 Feb 21;17:100544. doi: 10.1016/j.conctc.2020.100544. eCollection 2020 Mar. PMID 32154430
- [Background] Peng KP, Chiou JF, Chen YT, Liu TZ. Is the blood donated by habitual nut quid chewers suitable for use in transfusion? J Formos Med Assoc. 2010 Feb;109(2):106-12. doi: 10.1016/S0929-6646(10)60030-7. PMID 20206834
- [Background] Raja M, Saha S, Mohd S, Narang R, Reddy LV, Kumari M. Cognitive Behavioural Therapy versus Basic Health Education for Tobacco Cessation among Tobacco Users: A Randomized Clinical Trail. J Clin Diagn Res. 2014 Apr;8(4):ZC47-9. doi: 10.7860/JCDR/2014/8015.4279. Epub 2014 Apr 15. PMID 24959516
- [Background] Senn M, Baiwog F, Winmai J, Mueller I, Rogerson S, Senn N. Betel nut chewing during pregnancy, Madang province, Papua New Guinea. Drug Alcohol Depend. 2009 Nov 1;105(1-2):126-31. doi: 10.1016/j.drugalcdep.2009.06.021. Epub 2009 Aug 7. PMID 19665325
- [Background] Shirzaiy, M., & Neshat, F. (2020). Effect of areca nut on oral health: A review. Journal of Research in Dental and Maxillofacial Sciences, 5(3), 1-6.
- [Background] Siddiqi K, Dogar O, Rashid R, Jackson C, Kellar I, O'Neill N, Hassan M, Ahmed F, Irfan M, Thomson H, Khan J. Behaviour change intervention for smokeless tobacco cessation: its development, feasibility and fidelity testing in Pakistan and in the UK. BMC Public Health. 2016 Jun 10;16:501. doi: 10.1186/s12889-016-3177-8. PMID 27287429
- [Background] Song H, Wan Y, Xu YY. Betel quid chewing without tobacco: a meta-analysis of carcinogenic and precarcinogenic effects. Asia Pac J Public Health. 2015 Mar;27(2):NP47-57. doi: 10.1177/1010539513486921. Epub 2013 May 10. PMID 23666841
- [Background] Sotto PP, Mendez AJ, Herzog TA, Cruz C, Chennaux JSN, Legdesog C, Paulino YC. Barriers to Quitting Areca Nut Consumption and Joining a Cessation Program as Perceived by Chewer and Nonchewer Populations in Guam. Subst Use Misuse. 2020;55(6):947-953. doi: 10.1080/10826084.2020.1716012. Epub 2020 Jan 24. PMID 31973623
- [Background] Strickland SS, Duffield AE. Anthropometric status and resting metabolic rate in users of the areca nut and smokers of tobacco in rural Sarawak. Ann Hum Biol. 1997 Sep-Oct;24(5):453-74. doi: 10.1080/03014469700005212. PMID 9300122
- [Background] Strickland SS, Veena GV, Houghton PJ, Stanford SC, Kurpad AV. Areca nut, energy metabolism and hunger in Asian men. Ann Hum Biol. 2003 Jan-Feb;30(1):26-52. doi: 10.1080/03014460210157448. PMID 12519653
- [Background] Szumilas M. Explaining odds ratios. J Can Acad Child Adolesc Psychiatry. 2010 Aug;19(3):227-9. No abstract available. PMID 20842279
- [Background] Tahir ZH, Doss JG & Jaafar N. (2003). High-risk habits in relation to oral cancer in a Bajau community. [Master's thesis, Universiti Malaya]
- [Background] Taylor RF, al-Jarad N, John LM, Conroy DM, Barnes NC. Betel-nut chewing and asthma. Lancet. 1992 May 9;339(8802):1134-6. doi: 10.1016/0140-6736(92)90732-i. PMID 1349367
- [Background] Tham J, Sem G, Sit E, Tai MC. The ethics of betel nut consumption in Taiwan. J Med Ethics. 2017 Nov;43(11):739-740. doi: 10.1136/medethics-2016-103990. Epub 2017 Mar 6. PMID 28265049
- [Background] Tsai JF, Jeng JE, Chuang LY, Ho MS, Ko YC, Lin ZY, Hsieh MY, Chen SC, Chuang WL, Wang LY, Yu ML, Dai CY, Ho C. Habitual betel quid chewing as a risk factor for cirrhosis: a case-control study. Medicine (Baltimore). 2003 Sep;82(5):365-72. doi: 10.1097/01.md.0000090401.56130.59. PMID 14530785
- [Background] Warnakulasuriya S, Trivedy C, Peters TJ. Areca nut use: an independent risk factor for oral cancer. BMJ. 2002 Apr 6;324(7341):799-800. doi: 10.1136/bmj.324.7341.799. No abstract available. PMID 11934759
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- [Background] Winstock AR, Trivedy CR, Warnakulasuriya KA, Peters TJ. A dependency syndrome related to areca nut use: some medical and psychological aspects among areca nut users in the Gujarat community in the UK. Addict Biol. 2000 Apr 1;5(2):173-9. doi: 10.1080/13556210050003766. PMID 20575832
- [Background] Winstock A. Areca nut-abuse liability, dependence and public health. Addict Biol. 2002 Jan;7(1):133-8. doi: 10.1080/13556210120091509. PMID 11900633
- [Background] Wong, T. Y., Jin, Y. T., Chen, H. O., & Lin, L. M. (1992). Studies on Taiwan betel quid carcinogenicity in hamster cheek pouch. Chin Dent J, 11(4), 155-162.
- [Background] IARC Working Group on the Evaluation of Carcinogenic Risks to Humans. Betel-quid and areca-nut chewing and some areca-nut derived nitrosamines. IARC Monogr Eval Carcinog Risks Hum. 2004;85:1-334. No abstract available. PMID 15635762
- [Background] Yap SF, Ho PS, Kuo HC, Yang YH. Comparing factors affecting commencement and cessation of betel quid chewing behavior in Taiwanese adults. BMC Public Health. 2008 Jun 5;8:199. doi: 10.1186/1471-2458-8-199. PMID 18533044
- [Background] Yusoff MSB. (2019). ABC of content validation and content validity index calculation. Education in Medicine Journal, 11(2):49-54.
- [Background] Zain, R. B., Fukano, F., Razak, I. A., Shanmuhasuntharam, P., Ikeda, N., & Rahman, Z. A. A. (1999). Risk factors for oral leukoplakia: a comparison of two ethnic groups in Malaysia. Oral oncology, 6, 207-10.

DOCUMENTS (1):
  • Informed Consent Form (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT05782166/ICF_001.pdf